CLINICAL TRIAL: NCT05632367
Title: The Effects of Nutritional Characteristics of Obese Men and Women on Their Sexual Functions.
Brief Title: Relationship Between Nutrition and Sexual Activity
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Fulya Calikoglu, MD, PhD; Academician; Principle Investigator, Istanbul University
Other Study IDs: 2015/1100
Record Dates: First submitted 2022-11-13; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Sexual Dysfunction; Mediterranean Diet; Aphrodisiac Foods; Obesity; Healthy Eating Index
Keywords: SHIM; IEFF; Sexual Dysfunction; Aphrodisiac foods; Mediterranean Diet; Healthy Eating Index
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sexuality is integral to personality, influencing feelings, thoughts, actions, and physical and mental health. Female sexual dysfunction is a fairly common condition that covers four main areas: hypoactive sexual desire disorder, arousal disorder, orgasmic disorder, and sexual pain disorder. Although incidence and prevalence rates vary, it has been reported that women range between 30% and 50%.

Male sexual dysfunction is not a single disease. Male sexual arousal refers to the entire process of sexual activity for men, including penile erection, penile penetration, ejaculation, and any obstruction in a single connection. It is a significant psychological distress for affected men, their sexual partners, and their health-related quality of life. Sexual dysfunctions are common among men of all ages and ethnic and cultural backgrounds. It is reported in the literature that 52% of men between the ages of 40-70 experience various degrees of sexual dysfunction.

Cardiovascular disease, smoking, obesity, sedentary lifestyle, diabetes, hypertension, hyperlipidemia, and metabolic syndrome are risk factors for sexual dysfunction. Although the positive effects of adopting healthy lifestyle changes and dietary habits in reducing the risks of these diseases have been proven, few studies have evaluated the impact of these treatment approaches on sexual dysfunction.

Studies evaluating the relationship between diet and erectile dysfunction have focused more on men with diabetes. Some small studies have also shown that lifestyle modification and weight loss interventions improve erectile dysfunction in men with significant cardiovascular risks. The same is valid for female sexual dysfunction. The Western diet and its components are indirectly associated with sexual morbidity. The Western diet has processed foods, refined carbohydrates, and high sodium and monounsaturated fat content, which have been widely linked to the development of MetS, obesity, and diabetes. These comorbidities are also risk factors for female sexual dysfunction as well.

This study aims to evaluate the relationship between the eating habits of obese and non-obese men and women and their sexual functions.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with menstrual bleeding
2. Sexually active male and female patients
3. 18 years and older age

Exclusion Criteria:

1. <18 years of age
2. Female patients with menopause
3. Female patients that have undergone hormone therapy in the last 12 months
4. Sexually inactive male and female patients
5. Patients with diabetes
6. Patients with a history of psychiatric illness
7. Patients with cognitive impairment
8. Patients with hormone-dependent tumors
9. Patients taking a drug known to reduce sexual desire

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study was selected among adult obesity patients who were followed up and treated in the last six months of 2015 at Istanbul University Istanbul Medical Faculty Obesity Polyclinic. 185 patients aged 18 years and over were included in the study.
Sampling Method: Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Sexual function in obese women [ Time Frame: through study completion, an average of 6 months] | Based on The Female Sexual Function Index (FSFI) questionnaire
  A domain score of zero indicates that the subject reported having no sexual activity during the past month Desire: Score Range 1-5; Min-Max score 1.2-6.0 Arousal: Score Range 0-5; Min-Max score 0-6.0 Lubrication: Score Range 0-5; Min-Max score 0-6.0 Orgasm: Score Range 0 (or 1)-5; Min-Max score 0-6.0 Satisfaction: Score Range 0-5; Min-Max score 0.8-6.0 Pain: Score Range 0-5; Min-Max score 0-6.0
Sexual function in non-obese women [ Time Frame: through study completion, an average of 6 months] | Based on The Female Sexual Function Index (FSFI) questionnaire
  A domain score of zero indicates that the subject reported having no sexual activity during the past month Desire: Score Range 1-5; Min-Max score 1.2-6.0 Arousal: Score Range 0-5; Min-Max score 0-6.0 Lubrication: Score Range 0-5; Min-Max score 0-6.0 Orgasm: Score Range 0 (or 1)-5; Min-Max score 0-6.0 Satisfaction: Score Range 0-5; Min-Max score 0.8-6.0 Pain: Score Range 0-5; Min-Max score 0-6.0
Sexual function in obese men [ Time Frame: through study completion, an average of 6 months] | Based on International Index of Erectile Function (IIEF) questionnaire
  The possible scores for the IIEF-5 range from 5 to 25, and ED was classified into five categories based on the scores: severe (5-7), moderate (8-11), mild to moderate (12-16), mild (17-21), and no ED (22-25).
Sexual function in non-obese men [ Time Frame: through study completion, an average of 6 months] | Based on International Index of Erectile Function (IIEF) questionnaire
  The possible scores for the IIEF-5 range from 5 to 25, and ED was classified into five categories based on the scores: severe (5-7), moderate (8-11), mild to moderate (12-16), mild (17-21), and no ED (22-25).
Evaluation of which nutrients the participants consume weekly [ Time Frame: through study completion, an average of 6 months] | Based on Mediterranean Diet Assessment Tool
  Mediterranean Diet Assessment Scale; It is a questionnaire consisting of 14 questions, including the type of essential oil used by the patients in meals, the amount of olive oil consumed daily, fruit and vegetable portions, margarine-butter and red meat consumption, weekly consumption of wine, pulses, fish-seafood, snacks, nuts, cake, olive oil tomato sauce consumption and whether white meat is preferred more than red meat. 1 or 0 points are taken for each question asked according to the amount of consumption, and the total score is calculated. A score of 7 and above indicates that the individual has an acceptable degree of adherence to the Mediterranean diet. A score of 9 and above shows that the individual strictly follows the Mediterranean diet.
Evaluation of which nutrients the participants consume weekly [ Time Frame: through study completion, an average of 6 months] | Based on Alternative Healthy Eating Index
  The AHEI grades the diet, assigning a score ranging from 0 (nonadherence) to 110 (perfect adherence), based on how often eat certain healthy and unhealthy foods.
  For example, someone who reports eating no daily vegetables would score a zero, while someone who ate five or more servings a day would earn a 10. For an unhealthy option, such as sugar-sweetened drinks or fruit juice, scoring is reversed: a person who eats one or more servings would score a zero, and zero servings would earn a 10.

REFERENCES:
- [Result] Esposito K, Ciotola M, Giugliano F, De Sio M, Giugliano G, D'armiento M, Giugliano D. Mediterranean diet improves erectile function in subjects with the metabolic syndrome. Int J Impot Res. 2006 Jul-Aug;18(4):405-10. doi: 10.1038/sj.ijir.3901447. Epub 2006 Jan 5. PMID 16395320
- [Result] La J, Roberts NH, Yafi FA. Diet and Men's Sexual Health. Sex Med Rev. 2018 Jan;6(1):54-68. doi: 10.1016/j.sxmr.2017.07.004. Epub 2017 Aug 1. PMID 28778698
- [Result] Srivatsav A, Balasubramanian A, Pathak UI, Rivera-Mirabal J, Thirumavalavan N, Hotaling JM, Lipshultz LI, Pastuszak AW. Efficacy and Safety of Common Ingredients in Aphrodisiacs Used for Erectile Dysfunction: A Review. Sex Med Rev. 2020 Jul;8(3):431-442. doi: 10.1016/j.sxmr.2020.01.001. Epub 2020 Mar 2. PMID 32139335
- [Result] Cassidy A, Franz M, Rimm EB. Dietary flavonoid intake and incidence of erectile dysfunction. Am J Clin Nutr. 2016 Feb;103(2):534-41. doi: 10.3945/ajcn.115.122010. Epub 2016 Jan 13. PMID 26762373
- [Result] Mykoniatis I, Grammatikopoulou MG, Bouras E, Karampasi E, Tsionga A, Kogias A, Vakalopoulos I, Haidich AB, Chourdakis M. Sexual Dysfunction Among Young Men: Overview of Dietary Components Associated With Erectile Dysfunction. J Sex Med. 2018 Feb;15(2):176-182. doi: 10.1016/j.jsxm.2017.12.008. Epub 2018 Jan 8. PMID 29325831
- [Result] Weinberger JM, Houman J, Caron AT, Anger J. Female Sexual Dysfunction: A Systematic Review of Outcomes Across Various Treatment Modalities. Sex Med Rev. 2019 Apr;7(2):223-250. doi: 10.1016/j.sxmr.2017.12.004. Epub 2018 Feb 3. PMID 29402732
- [Result] Towe M, La J, El-Khatib F, Roberts N, Yafi FA, Rubin R. Diet and Female Sexual Health. Sex Med Rev. 2020 Apr;8(2):256-264. doi: 10.1016/j.sxmr.2019.08.004. Epub 2019 Oct 25. PMID 31669123